CLINICAL TRIAL: NCT00700947
Title: Beta-Blockade in Chronic Mitral Regurgitation: Moving From the Laboratory Experiment to Clinical Investigation
Brief Title: Using Beta Blockers to Treat Mitral Regurgitation
Acronym: REGURG
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding terminated
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007H0120; AHA-0335098N (Other: American Heart Association)
Record Dates: First submitted 2007-12-26; First posted 2008-06-19 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Heart Disease; Mitral Regurgitation; Heart Valve Disease; Mitral Valve Insufficiency
Keywords: Heart Disease; Mitral Regurgitation; Heart Valve Disease; Mitral Valve Insufficiency; Heart Surgery; Heart Valve Surgery
MeSH Terms: conditions — Heart Diseases; Mitral Valve Insufficiency; Heart Valve Diseases | interventions — Adrenergic beta-Antagonists; Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1 (Experimental): Patients who are asymptomatic with normal left ventricular systolic function and who agree to be treated medically for severe primary mitral regurgitation with Beta-blocker therapy. Patients may entered into the Arm 2 (surgical treatment) later on when they develop symptoms or enlarged left ventricle or left ventricular dysfunction or wishes to have surgical treatment of severe primary mitral regurgitation.
  Interventions: Drug: Beta-blocker therapy (TOPROL-XL® )
- 2 (No Intervention): Patients will be surgically treated for severe primary mitral regurgitation as a routine clinical care if they want to be treated surgically or develop symptoms or significant adverse left ventricular remodeling or left ventricular dysfunction.
- 3 (No Intervention): Health Control includes the subjects with no remarkable past medical history and not currently taking any medications. Normal subjects will be used for comparison with patients with severe primary mitral regurgitation in term of clinical, echocardiographic and neuro-hormonal findings.

INTERVENTIONS:
Drug: Beta-blocker therapy (TOPROL-XL® ) — Patients who are asymptomatic with normal left ventricular systolic function and wish to be medically treated for severe primary mitral regurgitation with Beta-blocker.
  Arms: 1

SUMMARY:
The purpose of this study tests whether beta-blocker will benefit asymptomatic patients with chronic primary mitral regurgitation.

DETAILED DESCRIPTION:
The purpose of this study tests 1) whether Toprol xl, a beta-blocker will benefit asymptomatic patients with chronic primary mitral regurgitation; 2) investigate the effects of chronic mitral regurgitation on left ventricular remodeling, left ventricular function,exercise capacity and clinical symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sever primary mitral regurgitation
* Normal subjects

Exclusion Criteria:

* Left ventricle ejection fraction of <55% pre and post operation
* Pregnancy or Lactation
* Secondary mitral regurgitation due to coronary artery disease, cardiomyopathy, uncontrolled hypertension, or severe aortic stenosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-10 (Actual); Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Change on Neurohormonal Measurements | Baseline, 6 months
  Change is calculated as the value at 6 months minus the value at baseline. The following neurohormones are measured: Brain type Natriuretic Peptide (BNP), tumor necrosis factor- alpha ( TNF- alpha), norepinephrine, epinephrine and plasma renin activity.
Change in Left Ventricular Ejection Fraction | Baseline, 6 months
  Measured on Echocardiogram. Change is calculated as the value at 6 months minus the value at baseline. Assess the systolic function.
Change on Left Ventricle end- Diastolic (LVEDD) and end-Systolic dimensions | Baseline, 6 months
  Measured on Echocardiogram. Change is calculated as the value at 6 months minus the value at baseline. Assess Left ventricular remodeling
Change on Left Ventricle end- Diastolic (LVEDD) and end-Systolic Volumes | Baseline, 6 months
  Measured on Echocardiogram. Change is calculated as the value at 6 months minus the value at baseline. Assess Left ventricular remodeling
Change on Left Ventricular Mass | Baseline, 6 months
  Measured on Echocardiogram. Change is calculated as the value at 6 months minus the value at baseline. Assess Left ventricular remodeling

SECONDARY OUTCOMES:
Change on the Regurgitant Stroke Volume | 6 months
  Measured on Echocardiogram. This will be calculated using the proximal isovelocity surface area (PISA) method.Change is calculated as the value at 6 months minus the value at baseline.
Change in Pulmonary Venous Systolic Flow Reversal | Baseline, 6 months
  Measured on Echocardiogram Color Doppler mapping of Mitral Regurgitation (MR) jets will be used to semiquantitative asses severity of MR using a 4 point scale( 1-4, where higher scores denotes worse outcomes).

CONTACTS AND LOCATIONS:
Overall Officials: Min Pu, MD, Principal Investigator — The Wake Forest University
Locations (1):
- Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
We currently have no plan to share participant data.

REFERENCES:
- [Background] Yang H, Davidson WR Jr, Chambers CE, Pae WE, Sun B, Campbell DB, Pu M. Preoperative pulmonary hypertension is associated with postoperative left ventricular dysfunction in chronic organic mitral regurgitation: an echocardiographic and hemodynamic study. J Am Soc Echocardiogr. 2006 Aug;19(8):1051-5. doi: 10.1016/j.echo.2006.03.016. PMID 16880102
- [Background] Pu M, Gao Z, Li J, Sinoway L, Davidson WR Jr. Development of a new animal model of chronic mitral regurgitation in rats under transesophageal echocardiographic guidance. J Am Soc Echocardiogr. 2005 May;18(5):468-74. doi: 10.1016/j.echo.2004.10.005. PMID 15891757
- [Result] Pu M, Gao Z, Pu DK, Davidson WR Jr. Effects of early, late, and long-term nonselective beta-blockade on left ventricular remodeling, function, and survival in chronic organic mitral regurgitation. Circ Heart Fail. 2013 Jul;6(4):756-62. doi: 10.1161/CIRCHEARTFAILURE.112.000196. Epub 2013 Apr 11. PMID 23580745
- [Result] Pu M, Gao Z, Zhang X, Liao D, Pu DK, Brennan T, Davidson WR Jr. Impact of mitral regurgitation on left ventricular anatomic and molecular remodeling and systolic function: implication for outcome. Am J Physiol Heart Circ Physiol. 2009 Jun;296(6):H1727-32. doi: 10.1152/ajpheart.00882.2008. Epub 2009 Mar 27. PMID 19329766
- [Result] Pu M. The frequency, impact, and management of mitral regurgitation in patients with heart failure. Curr Cardiol Rep. 2006 May;8(3):226-31. doi: 10.1007/s11886-006-0038-6. PMID 17543250